CLINICAL TRIAL: NCT01170988
Title: Comparison of Coronary Flow Reserve in Two Different Bypass Techniques (T-graft Technique Versus Isolated Graft Technique) Using Magnetic Resonance Technology (MRT)
Brief Title: Coronary Flow Rate Measurement in T-Grafts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Collaborators: Bethanien Krankenhaus gGmbH (Other)
Responsible Party: Principal Investigator, Arndt-H. Kiessling, Head cardiovascular research, Johann Wolfgang Goethe University Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FLUSS001AHK
Record Dates: First submitted 2010-07-27; First posted 2010-07-28 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Coronary Heart Disease
Keywords: patients scheduled for bypass grafting
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- surgical procedure (Other): T-graft bypass or conventional bypass
  Interventions: Procedure: T-Graft

INTERVENTIONS:
Procedure: T-Graft — T-Graft

SUMMARY:
Is the surgical treatment of patients with coronary heart disease using the T-graft technique an adequate solution that provides a sufficient myocardial flow reserve? A magnetic resonance examination (MRI) is required.

ELIGIBILITY:
Inclusion Criteria:

* coronary heart disease
* Age > 18 ys
* Ejection fraction > 45%

Exclusion Criteria:

* myocardial infarction
* Re-Intervention

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Coronary flow reserve | within 4-6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Johann Wolfgang Goethe Universitätsklinikum, Frankfurt am Main, Germany